CLINICAL TRIAL: NCT01279070
Title: Efficacy of Repyflec Cognitive Remediation Group Training in Cognition, Functional Outcomes and Psychiatric Symptoms of Outpatients With Schizophrenia.
Brief Title: Efficacy of Repyflec Cognitive Remediation Group Training in Schizophrenia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fundació Sant Joan de Déu (Other)
Responsible Party: Principal Investigator, Aida Farreny, Dr. Aida Farreny, Fundació Sant Joan de Déu
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REPYFLEC Clinical Trial
Record Dates: First submitted 2011-01-14; First posted 2011-01-19 (Estimated); Results first posted 2013-08-15 (Estimated); Last update posted 2013-08-23 (Estimated); Status verified 2013-05

CONDITIONS: Indication for Modification of Patient Cognitive Status
Keywords: Schizophrenia; Cognitive remediation; Group training; Executive function; Social functioning
MeSH Terms: conditions — Schizophrenia; Social Adjustment | interventions — Cognitive Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- REPYFLEC cognitive remediation training (Experimental): REPYFLEC cognitive remediation as a Problem solving and Cognitive flexibility group training.
  Interventions: Behavioral: Repyflec cognitive remediation training
- Leisure group (Active Comparator): Leisure group is a stimulating activity focused on socialization through group dynamics, board games, "coffee and talk".
  Interventions: Behavioral: Repyflec cognitive remediation training

INTERVENTIONS:
Behavioral: Repyflec cognitive remediation training — Comparison of 32 Repyflec group sessions among 32 leisure group sessions where we stimulated non-specific cognitive perform.
  Other Names: Cognitive remediation therapy; Cognitive rehabilitation; Cognitive training

SUMMARY:
The purpose of this study was to develop an integrative intervention for schizophrenia taking into account previous efficacious therapies. Thus, our aim was to evaluate the efficacy of our cognitive remediation group training: Problem Solving and Cognitive Flexibility training (REPYFLEC), focused to improve neurocognition and functioning in schizophrenia patients. We hypothesized that training executive function and metacognition would allow us to achieve improvements in neurocognition, functioning and psychiatric symptoms of patients with schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of schizophrenia or schizoaffective disorder
* More than 2 years illness duration
* Literate
* Mini Mental Status Examination score over 24
* Global Assessment of Functioning scores between 40 and 70

Exclusion Criteria:

* Current acute illness exacerbation
* Mental Retardation
* Neurological disorder which impairs cognition
* Currently participating in social skills training or cognitive remediation
* Change of antipsychotic medication one month before the trial or during the 40 study weeks
* Diagnosis of alcohol or drug dependence within 6 months of trial commencement.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2006-09; Primary Completion 2009-01 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aida Farreny, PhD Psycho., Principal Investigator — Fundació Sant Joan de Déu
Locations (1):
- Parc Sanitari Sant Joan de Déu, Sant Boi de Llobregat, Barcelona, Spain

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment started on January 2007 and finished on May 2010. We have worked in different outpatient Rehabilitation Centers and we incorporated experimental and control group as a part of their rehabilitation planning. We have worked in 6 different centers.
Groups:
- Experimental Group (Repyflec Cognitive Remediation): Cognitive remediation (CR) group training (Repyflec)
  REPYFLEC CR is a strategy-based training that targets executive function and metacognition. It is carried out using paper and pencil and a blackboard (required to develop some of the tasks, explanations,examples, etc.); in a group format (4-6 participants), over 4 months twice a week and consisting of 32 sessions lasting 1 h. We developed a Spanish manual where training is described session by session; incorporating the materials for developing sessions, some theoretical points and bibliography for therapists. Working contents are divided into two main areas: Problem Solving (PS) and Cognitive Flexibility (CF).
- Leisure Group (Control Group): Leisure group
  Parallel to the experimental group, a leisure control group was established which participated in 32 stimulating and socializing activities (e.g., card games, board games, "coffee & talk", etc.) over 4 months twice a week and lasting 1 h.
Period: Overall Study
Arm/Group | Experimental Group (Repyflec Cognitive Remediation) | Leisure Group (Control Group)
Started | 34 (34 outpatients were randomly assigned to 32 sessions of REPYFLEC.) | 28 (28 outpatients were randomly assigned to 32 sessions of leisure group.)
Completed | 29 (5 outpatients left the treatment up to 2 months after starting REPYFLEC.) | 24 (4 outpatients left the leisure group up to 2 months after starting Leisure group.)
Not Completed | 5 | 4
Not completed — Withdrawal by Subject | 2 | 3
Not completed — Acute exacerbation | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Leisure Group: Leisure group has got same number of sessions and timing than experimental group
- Repyflec Training: Cognitive remediation treatment
- Total: Total of all reporting groups
Arm/Group | Leisure Group | Repyflec Training | Total
Number analyzed (Participants) | 28 | 34 | 62
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 28 | 34 | 62
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 41.9 (6.7) | 39.6 (8.2) | 40.6 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 11 | 20
  Male | 19 | 23 | 42
Region of Enrollment [Number; unit: participants]
  Spain | 28 | 34 | 62

OUTCOME MEASURES:

1. Primary Outcome: Executive Function
Description: Behavioral Assessment of the Dysexecutive Syndrome (BADS). This scale evaluates cognitive flexibility, inhibition of impulsive responses, planning and organization, working memory and time-estimation capacity. All subscales (Rule shift cards, Action Program, Key search, Temporal judgment, Zoo map and Six elements) were administered. We used subscales raw scores which run from 0 to 4. The subscales' raw score is summarized and converted to standardized total score which run (min.
  12-max. 129). A higher score indicates better performance.
Time Frame: Change from baseline in executive function at 16 weeks (post-treatment)
Population: The sample size required was calculated according to the main study objective which consisted of achieving an improvement in social functioning according to the Living Skills Profile (LSP) scale. It was estimated that a sample of 27 patients per group would have a power of 80% at a significance level of 5% to detect these differences.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- REPYFLEC Cognitive Remediation Group Training: REPYFLEC CR is a strategy-based training that targets executive function and metacognition. It is carried out using paper and pencil and a blackboard (required to develop some of the tasks, explanations, examples, etc.); in a group format (4-6 participants), over 4 months twice a week and consisting of 32 sessions lasting 1 h. We developed a Spanish manual where training is described session by session; incorporating the materials for developing sessions, some theoretical points and bibliography for therapists. Working contents are divided into two main areas: Problem Solving (PS) and Cognitive Flexibility (CF). In the PS module (16 sessions), training in executive function,thinking processes and self-monitoring was emphasized.In the CF module (16 sessions), all the tasks require practice of cognitive flexibility combined with other executive abilities such as planning or self-monitoring.
- Leisure & Socialization Group: The leisure group consists in 32 stimulating and socializing group activities (e.g., card games, board games, "coffee & talk", geography review, etc.)without specific goals.
Arm/Group | REPYFLEC Cognitive Remediation Group Training | Leisure & Socialization Group
Number analyzed (Participants) | 29 | 24
units on a scale
  BADS total standardized score (from 12 to 129) | 99.5 (14.5) | 95.7 (13.5)
  BADS Key search subscale (from 0 to 4) | 2.7 (1.2) | 1.7 (1.3)
Statistical Analysis 1: Comparison: REPYFLEC Cognitive Remediation Group Training vs Leisure & Socialization Group; To evaluate intervention efficacy on the BADS(Total score and Key search subtest),linear mixed-effects models were fitted using Restricted Maximum Likelihood (REML.An unstructured correlation matrix was used to account for correlation among several observations for each subject.The dependent variable comprised the measures at 16 weeks while the baseline value of the BADS,intervention group(REPYFLEC group vs Leisure group),time and the interaction term (time×treatment)were included as covariates; Test type: Superiority or Other; p < 0.05, Mixed Models Analysis; Effect size = 0.43, 95% CI 2-sided [0.1 to 0.7] — In all the models,adjusted mean difference between the two groups,standardized treatment effect (ES) and confidence intervals were calculated.All the estimates obtained with these models remain unbiased under the missing at random (MAR)assumption

2. Primary Outcome: Executive Function
Description: Behavioral Assessment of the Dysexecutive Syndrome (BADS) (Wilson et al., 1996). This scale evaluates cognitive flexibility, inhibition of impulsive responses, planning and organization, working memory and time-estimation capacity. All subscales (Rule shift cards, Action Program, Key search, Temporal judgement, Zoo map and Six elements) were administered. We used subscales raw scores which run from 0 to 4. The subscales' raw score is summarized and converted to standardized total score which run (min.
  12-max. 129). A higher score indicates better performance.
Time Frame: Change from baseline in executive functioning at 40 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- REPYFLEC Cognitive Group Trainining: REPYFLEC is a strategy-based training, explicitly described from session to session, which is carried out using pencil and paper with a blackboard as visual support. This format allows results to be replicated with rigour. The working content is divided into two principal areas: Problem solving (PS) and Cognitive Flexibility (CF). In the PS block, training in executive function, the thinking process and self-monitoring was emphasized. In the CF block, the tasks require the use of cognitive flexibility for successful completion. Some activities seek to promote training of other functions such as memory, working memory, sustained attention and language. Development of training was performed taking into account the contextual bases of learning, mainly using techniques as "modelling" to foster coping abilities, "molding", "self-monitoring", "errorless learning" and "Socratic questioning". REPYFLEC is carried out in a group format (4-6), consisting of 32 sessions lasting 1 hour.
- Leisure & Socialization Group: Parallel to the experimental group, a leisure group was established (control group) which participated in 32 stimulating and socializing activities (e.g., card games, board games, "coffee & talk", geography review, etc).
Arm/Group | REPYFLEC Cognitive Group Trainining | Leisure & Socialization Group
Number analyzed (Participants) | 28 | 19
units on a scale
  BADS standardized total score (min.12-max.129) | 101.8 (10.1) | 94.5 (14.7)
  BADS Key search subscale (from 0 to 4) | 3 (1.1) | 1.7 (1.4)
Statistical Analysis 1: Comparison: REPYFLEC Cognitive Group Trainining vs Leisure & Socialization Group; To evaluate intervention efficacy on the BADS(Total score and Key search subtest),linear mixed-effects models were fitted using Restricted Maximum Likelihood(REML).An unstructured correlation matrix was used to account for correlation among several observations for each subject.The dependent variable comprised the measures at 40 weeks while the baseline value of the BADS,intervention group(REPYFLEC group vs Leisure group),time and the interaction term (time×treatment)were included as covariates; Test type: Superiority or Other; p < 0.05, Mixed Models Analysis; Effect Size = 0.42, 95% CI 2-sided [0.1 to 0.7] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Psychosocial Functioning
Description: The Spanish validation of the Life Skills Profile (LSP)was used. This scale measures functionality in daily life activities such as self-care, social behavior and autonomy. Raw scoring was used for the various subscales which are summarized for the total (min. 39-max. 156) with a higher score indicating a better result.
  The 5 subscales are: Self-care, Non-turbulence, Social contact, Communication and Responsibility. We used the Spanish validation of the Social Functioning Scale (SFS)for measuring social behavior and relationships, autonomy, employment-occupation and leisure. Raw scoring was used for each subscale and for total score (min. 0-max. 223) with a higher score indicating a better result. All 7 subscales were administered: social engagement/ withdrawal, interpersonal behavior, independence-competence, independence-performance, pro-social activities, recreation and employment/ occupation.
Time Frame: Change from baseline in social functioning scales at 16 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Repyflec Training | Leisure Group
Number analyzed (Participants) | 29 | 24
units on a scale
  LSP Total Score (min. 39-max. 156) | 137.4 (6.9) | 133.6 (11.4)
  SFS Total Score (min. 0-max. 223) | 108.8 (17.6) | 105.9 (19.3)
Statistical Analysis 1: Comparison: Repyflec Training vs Leisure Group; To evaluate intervention efficacy on the LSP, linear mixed-effects models were fitted using Restricted Maximum Likelihood (REML). An unstructured correlation matrix was used to account for correlation among several observations for each subject. The dependent variable comprised the measures at 16 weeks while the baseline value of the LSP, intervention group (REPYFLEC group vs Leisure group), time and the interaction term (time×treatment) were included as covariates; Test type: Superiority or Other; p < 0.05, Mixed Models Analysis; Effect Size = 0.33, 95% CI 2-sided [0.06 to 0.6] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Psychosocial Functioning
Description: as for outcome 3
Time Frame: Change from baseline in social functioning scales at 40 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Repyflec Training | Leisure Group
Number analyzed (Participants) | 28 | 19
units on a scale
  LSP Total Score (min. 39-max. 156) | 135.7 (7.7) | 132.9 (12)
  SFS Total Score (min. 0-max. 223) | 107 (16.6) | 107.2 (14.8)
Statistical Analysis 1: Comparison: Repyflec Training vs Leisure Group; To evaluate intervention efficacy on the LSP, linear mixed-effects models were fitted using Restricted Maximum Likelihood (REML). An unstructured correlation matrix was used to account for correlation among several observations for each subject. The dependent variable comprised the measures at 40 weeks while the baseline value of the LSP, intervention group (REPYFLEC group vs Leisure group), time and the interaction term (time×treatment) were included as covariates; Test type: Superiority or Other; p < 0.05, Mixed Models Analysis; Effect Size = 0.35, 95% CI 2-sided [0.09 to 0.6] — [estimate comment as in outcome 1, analysis 1]

5. Secondary Outcome: Psychiatric Symptoms
Description: The Spanish validation of the Positive and Negative Syndrome Scale (PANSS) was used for measuring positive, negative and general symptomatology. Total raw scoring obtained through the sum of the raw scores for each subscale was considered (min. 30-max. 210) with a score of 30 representing an absence of psychiatric symptoms.
Time Frame: Change from baseline in psychiatric symptoms scales at 16 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Repyflec Training | Leisure Group
Number analyzed (Participants) | 29 | 24
units on a scale
  Positive (from 7 to 49) | 11.5 (2.9) | 12.8 (3.5)
  Negative (from 7 to 49) | 16.6 (4.1) | 17.5 (5.2)
  General Psychopathology (from 16 to 112) | 27.5 (6) | 30.1 (6.1)
  PANSS Total score (min. 30-max. 210) | 55.6 (10.6) | 60.4 (12.3)
Statistical Analysis 1: Comparison: Repyflec Training vs Leisure Group; To evaluate intervention efficacy on the PANSS, linear mixed-effects models were fitted using Restricted Maximum Likelihood (REML). An unstructured correlation matrix was used to account for correlation among several observations for each subject. The dependent variable comprised the measures at 16 weeks while the baseline value of the PANSS, intervention group (REPYFLEC group vs Leisure group), time and the interaction term (time×treatment) were included as covariates; Test type: Superiority or Other; p < 0.05, Mixed Models Analysis; Effect Size = 0.3, 95% CI 2-sided [0.01 to 0.7] — [estimate comment as in outcome 1, analysis 1]

6. Secondary Outcome: Psychiatric Symptoms
Description: as for outcome 5
Time Frame: Change from baseline in psychiatric symptoms scales at 40 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Repyflec Training | Leisure Group
Number analyzed (Participants) | 28 | 19
units on a scale
  Positive (from 7 to 49) | 12.9 (3.3) | 14 (4.8)
  Negative (from 7 to 49) | 17.6 (3.7) | 16.9 (3.8)
  General Psychopathology (from 16 to 112) | 30.8 (5.7) | 30.8 (5)
  PANSS Total score (min. 30- max. 210) | 61.4 (9.5) | 61.8 (10.5)
Statistical Analysis 1: Comparison: Repyflec Training vs Leisure Group; To evaluate intervention efficacy on the PANSS, linear mixed-effects models were fitted using Restricted Maximum Likelihood (REML). An unstructured correlation matrix was used to account for correlation among several observations for each subject. The dependent variable comprised the measures at 40 weeks while the baseline value of the PANSS, intervention group (REPYFLEC group vs Leisure group), time and the interaction term (time×treatment) were included as covariates; Test type: Superiority or Other; p < 0.05, Mixed Models Analysis; Effect Size = 0.3, 95% CI 2-sided [0.01 to 0.7] — In all the models,adjusted mean difference between the two groups, standardized treatment effect (ES) and confidence intervals were calculated.All the estimates obtained with these models remain unbiased under the missing at random (MAR) assumption

ADVERSE EVENTS:
Time Frame: At baseline (week 0), post-treatment (week 16) and follow-up assessments (week 40). Two times per week during 16 weeks of intervention groups.
Description: There are not expected risks for the testing,interviews or REPYFLEC and control groups.However,there is the possibility that patients could get tired or feel a bit uncomfortable after completing groups or assessments.At interviews and cognitive testing there will be the option of taking short breaks to avoid fatigue and potential discomfort.
Groups:
- Leisure Group: Stimulating activities without specific goals and focused on leisure
- Repyflec Training: Cognitive remediation group treatment based on Problem Solving and Cognitive Flexibility
Arm/Group | Leisure Group | Repyflec Training
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/29
Other Adverse Events (participants affected / at risk) | 0/24 | 0/29

LIMITATIONS AND CAVEATS:
It would be useful to widen the assessment of cognitive measures and negative symptoms. Metacognition has not been appropriately studied.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No